CLINICAL TRIAL: NCT02266524
Title: Pharmacokinetics, Safety and Tolerability of Single Oral Doses (0.1, 0.2, 0.4 and 0.8 mg) of Tamsulosin Hydrochloride in Children With Voiding Disorders
Brief Title: Pharmacokinetics, Safety and Tolerability of Tamsulosin Hydrochloride in Children With Voiding Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 527.49
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Urination Disorders
MeSH Terms: conditions — Urination Disorders | interventions — Tamsulosin

ARMS (4):
- Tamsulosin hydrochloride, very low dose (Experimental)
  Interventions: Drug: Tamsulosin hydrochloride, very low dose
- Tamsulosin hydrochloride, low dose (Experimental)
  Interventions: Drug: Tamsulosin hydrochloride, low dose
- Tamsulosin hydrochloride, medium dose (Experimental)
  Interventions: Drug: Tamsulosin hydrochloride, medium dose
- Tamsulosin hydrochloride, high dose (Experimental)
  Interventions: Drug: Tamsulosin hydrochloride, high dose

INTERVENTIONS:
Drug: Tamsulosin hydrochloride, very low dose
  Other Names: Flomax®
  Arms: Tamsulosin hydrochloride, very low dose
Drug: Tamsulosin hydrochloride, low dose
  Other Names: Flomax®
  Arms: Tamsulosin hydrochloride, low dose
Drug: Tamsulosin hydrochloride, medium dose
  Other Names: Flomax®
  Arms: Tamsulosin hydrochloride, medium dose
Drug: Tamsulosin hydrochloride, high dose
  Other Names: Flomax®
  Arms: Tamsulosin hydrochloride, high dose

SUMMARY:
To investigate pharmacokinetics, safety, and tolerability of tamsulosin hydrochloride in children with voiding disorders

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls with (or a history of) voiding disorders
* Age: 5 to 15 years
* Body weight and height ≥ 5 % and ≤95 % of normal using nomograms
* Signed and dated written informed consent by the parent or guardian and, where appropriate, informed assent by the child, prior to admission into the study in accordance with good clinical practice (GCP) and the local legislation, has been obtained

Exclusion Criteria:

* Clinically significant abnormalities found at, or before randomization at Visit 2 [i.e., abnormal: vital signs (e.g., hypotension), ECGs, as well as significant findings during the physical examination], as determined by the investigator
* Clinically relevant conditions including, but not limited to, the following: gastrointestinal, cardiovascular (e.g., subjects that fall above the 90th percentile according to the blood pressure nomogram in the ISF), hepatic, renal, hematologic, metabolic (including diabetes mellitus), immunological, hormonal disorders, respiratory disease or cancer
* Subjects who had surgery within the last 30 days
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Subjects that have a neurological impairment or psychiatric disorder that prevents their comprehension of consent and their ability to comply with the protocol
* History of relevant orthostatic hypotension, fainting spells or blackouts. Postdural symptoms occurring (e.g., lightheadedness, dizziness, and fainting) with or without a change in blood pressure and / or pulse rate within 6 weeks of Visit 2
* Relevant acute infections, especially with regards to urinary tract infections or active genitourinary infection
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Subjects with known hypersensitivity to FLOMAX® (tamsulosin hydrochloride) or other alpha-blockers
* Use of medications classified as cytochrome P450 3A4 (CYP3A4) inhibitors and inducers within 10 days prior to administration of trial drug
* Intake of drugs with a long half-life (> 24 hours) within less than 10 half-lives of the respective drug prior to administration
* Participation in another trial with an investigational drug within 1 month prior to administration or during the trial
* Inability to comply with dietary regimen of study center
* Pregnancy or subjects that are breast feeding
* All subjects parents and guardians in the investigator's opinion who cannot understand the terms of the informed consent form and subject information

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | Up to 26 hours after drug administration
Time from dosing to maximum concentration of the analyte in plasma (tmax) | Up to 26 hours after drug administration
Area under the concentration-time curve of the analyte in plasma (AUC) | Up to 26 hours after drug administration
Percentage of the AUC0-∞ that is obtained by extrapolation (%AUCtz-∞) | Up to 26 hours after drug administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single-dose administration (AUC0-∞)
Terminal rate constant of the analyte in plasma (λz) | Up to 26 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 26 hours after drug administration
Mean residence time of the analyte in the body after po administration (MRTpo) | Up to 26 hours after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | Up to 26 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | Up to 26 hours after drug administration
Weight-normalized Cmax | Up to 26 hours after drug administration
Weight-normalized AUC0-∞ | Up to 26 hours after drug administration
Weight-normalized (AUC0-tz) | Up to 26 hours after drug administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration after single-dose administration (AUC0-tz)

SECONDARY OUTCOMES:
Number of patients with clinically relevant changes in physical examination | Pre-dose, up to 26 hours after drug administration
Number of patients with clinically relevant changes in vital signs (blood pressure, pulse rate, respiratory rate) | Pre-dose, up to 26 hours after drug administration
Number of patients with clinically relevant changes from baseline in orthostatic test | Pre-dose and 4 hours after drug administration
Number of patients with clinically relevant changes in 12-lead ECG | Pre-dose, up to 26 hours after drug administration
Number of patients with clinically relevant changes from baseline in laboratory tests | Pre-dose and 26 hours after drug administration
Number of patients with adverse events | Up to 7 days after drug administration
Global assessment of tolerability by the investigator on a 5-point rating scale | 26 hours after drug administration